CLINICAL TRIAL: NCT02899130
Title: Antiviral Effect of 3 Herbs in Chronic Inactive Carriers of Hepatitis B Virus. - A Randomized Placebo Controlled Clinical Trial
Brief Title: Effect of Polyherbal Formulation in Chronic Inactive Carriers of Hepatitis B Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OI- 002- 2016
Record Dates: First submitted 2016-09-08; First posted 2016-09-14 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyherbal (Experimental): Combination of 3 whole herbs in a capsule
  Interventions: Drug: Polyherbal
- Matching placebo (Placebo Comparator): Similar looking inert capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyherbal — Each capsule contains 3 herbs. Phyllanthus niruri, Boerhaavia diffusa, picrorhiza kurroa
  Other Names: Liver Kidney Care
  Arms: Polyherbal
Drug: Placebo — Inactive compound that is similar looking as the intervention
  Arms: Matching placebo

SUMMARY:
This trial will study the effect of a polyherbal capsule in lowering the viral load of patients with chronic Hepatitis B infection and record the incidence of from Hepatitis B surface antigen elimination in 12 months

DETAILED DESCRIPTION:
A placebo controlled randomised trial. 3 herbs that have proven effect on eliminating the virus and normalizing liver function will be given. Equally matched placebo (blinded) will be given randomly to patients. All parameters of hepatitis B infection will be compared between the randomized groups

ELIGIBILITY:
Inclusion Criteria:

* Adults aged above 18 years of age, with inactive chronic hepatitis B (HB) or immune tolerant phase, with or without dyslipidaemia and having all of the following

  1. HBsAg +ve for >6 months and anti-HBs negative
  2. Alanine amino transferase ≤ 2 upper limit of normal
  3. HBeAg positive or negative irrespective of viral DNA load
  4. Not currently on antiviral therapy for Chronic hepatitis B

Exclusion Criteria:

* Any one of the following

  1. Patients with decompensated liver disease of any etiology(characterized by elevated bilirubin, raised International normalized ratio, or a history of ascites, variceal hemorrhage,hepatic encephalopathy, Spontaneous bacterial peritonitis, hepatorenal syndrome or Hepatocellular carcinoma)
  2. Family history of hepatocellular carcinoma
  3. Patients with HIV and Hepatitis C virus co-morbidity
  4. Pregnant, attempting to conceive, or lactating women
  5. Patients with diabetes mellitus
  6. Recent history of acute coronary syndrome (<6months) or chronic coronary artery disease with poor left ventricular function (by physician / cardiology opinion)
  7. Patients with renal failure ( Creatinine clearance less than 60 ml/min)
  8. Active substance or alcohol abuse and concurrent use of corticosteroids or immunosuppressive agents.
  9. Presence of extra hepatic manifestations
  10. Previously treated with pegylated interferon within the last 2 years
  11. Positive fibroscan or ultrasound elastography showing evidence of fibrosis (F3 and above)
  12. Current or former employees of organic India
  13. Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.
  14. Refusing consent or physician uncomfortable with patient compliance to treatments or follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with change in mean Hepatitis B Virus (HBV) DNA by at least 2log10 units from baseline at end of treatment for those with HBV DNA ≥ 1000 IU/ml. | 12 months

SECONDARY OUTCOMES:
Number of patients with change in hepatitis B surface antigen titers from baseline for those with HBV DNA <1000 IU/ml | 12 months
Number of patients with Incidence of seroconversion from Hepatitis B surface antigen to anti-Hepatitis B surface antibody | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alben Sigamani, MD, Principal Investigator — Narayana Hrudayalaya Hospital
Locations (1):
- Mazumdar Shaw Mutispeciality Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided